CLINICAL TRIAL: NCT05791968
Title: Effects of a Standard Blood Bank Donation on Insulin Sensitivity in Adults With Pre-diabetes and Abdominal Obesity
Brief Title: Blood Donation Could Improve Insulin Sensitivity
Acronym: GLUCFER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Collaborators: SESCAM Centro Regional de Transfusión Toledo-Guadalajara. (Unknown)
Responsible Party: Principal Investigator, Ricardo Mora, Director of Exercise Physiology Laboratory, University of Castilla-La Mancha
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEIC-CHUT-969
Record Dates: First submitted 2023-03-17; First posted 2023-03-30 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2023-03

CONDITIONS: Ferritin; Insulin Sensitivity; Blood Donation
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Randomized, control group, trial (RCT)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: participants in the control group will have the standard blood bank donation venipuncture, but no blood will be withdrawn (sham donation).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DONATION GROUP (Active Comparator): Participants will be measured before and after a standard blood bank donation (450 mL of whole blood withdrawal)
  Interventions: Procedure: Whole blood standard donation
- CONTROL GROUP (Sham Comparator): Participants will be measured before and after a sham blood donation (0 mL of whole blood withdrawal)
  Interventions: Procedure: Whole blood standard donation

INTERVENTIONS:
Procedure: Whole blood standard donation — Effects of a standard whole blood donation on iron stores and insulin sensitivity.

SUMMARY:
Studies in the literature suggest that people with obesity have an excess of stored iron. There is possibly an inverse relationship between ferritin levels and the actions of insulin on glycemic control. The reduction of stored iron by simply donating blood could result in improvements in glycemic control in people with obesity and prediabetes. We propose, to reduce ferritin levels through a standard donation of a unit of whole blood, and to measure if it positively affects glycemic control.

DETAILED DESCRIPTION:
Individuals with pre-diabetes and abdominal obesity will be randomized to either a donation group (DON) or a control group (CONT) in a double-blind fashion (RCT).

Insulin sensitivity during an oral glucose tolerance test (OGTT) and isotopically measured rate of appearance of endogenous and exogenous glucose will be measured on 2 occasions.

1. Two weeks prior to DON/CONT
2. Two weeks after to DON/CONT

Indexes of the bodily iron stores will be measured after DON/CONT to evaluate if the primary treatment was effective.

ELIGIBILITY:
Inclusion Criteria:

* have not donated in the last 3 months
* IMC>25
* fasting blood glucose 100-125 mg/dL
* glycosylated hemoglobin levels between 5.7-6.4%

Exclusion Criteria:

* to not meet donor bank requirements
* insulin treatment for diabetes
* anemia
* hereditary hemochromatosis
* heart disease
* familial hypertriglyceridemia or hypobetalipoproteinemia
* any disease that requires medication that interferes with iron or glucose metabolism

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity during an oral glucose tolerance test (OGTT) | 7 months
  Measured with the calculations of Matsuda index
Ferritin blood level | 7 months
  iron stores index measured in blood
Turnover rate of endogenous and exogenous glucose | 7 months
  Measured using isotopic tracers.
Carbohydrate oxidation | 7 months
  Measured using indirect calorimetry
Continuous glucose monitoring | 7 months
  Interstitial blood glucose concentrations during 24-h

SECONDARY OUTCOMES:
Cuality of life | 7 months
  Measured by SF 12
Fasting lipid profile | 7 months
  blood analysis
Body composition (weight and body fat) | 7 months
  TANITA

CONTACTS AND LOCATIONS:
Locations (1):
- University of Castilla-La Mancha (Exercise Physiology Lab), Toledo, Toledo, Spain

IPD SHARING:
Plan to Share IPD: Undecided
data will be shared upon reasonable request.

REFERENCES:
- [Background] Moreno-Navarrete, J. M., M. Moreno, J. Puig, G. Blasco, F. Ortega, G. Xifra, W. Ricart and J. M. Fernandez-Real (2017).
- [Background] Van Pelt, D. W., S. A. Newsom, S. Schenk and J. F. Horowitz (2015).